CLINICAL TRIAL: NCT06840548
Title: A Phase I Study to Evaluate the Safety and Dosimetry of 68Ga-OncoCAIX in Patients With CAIX-positive Cancer
Brief Title: A Study to Evaluate the Safety and Dosimetry of 68Ga-OncoCAIX in Patients With CAIX-positive Cancer
Acronym: OncoCAIX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PH-CAIXGA-02/24; 2024-515607-19-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Clear Cell Renal Cell Carcinoma (ccRCC)
Keywords: clear cell renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: Patients are divided into two cohorts:
  * Cohort A: 3 female + 3 male patients without visceral or bone metastases, which would interfere with dosimetry evaluation of healthy organs.
  * Cohort B: all patients who meet the eligibility criteria (up to 14 patients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coort A (Experimental): 3 female + 3 male patients without visceral or bone metastases, which would interfere with dosimetry evaluation of healthy organs.
  Interventions: Drug: [68Ga]Ga-OncoCAIX
- Cohort B (Experimental): all patients who meet the eligibility criteria (up to 14 patients)
  Interventions: Drug: [68Ga]Ga-OncoCAIX

INTERVENTIONS:
Drug: [68Ga]Ga-OncoCAIX — Single intravenous bolus administration.

SUMMARY:
Phase I and multicenter study to evaluate the safety and dosimetry of 68Ga-OncoCAIX in patients with clear cell renal cell carcinoma.

DETAILED DESCRIPTION:
The Carbonic Anhydrase IX (CAIX) is a clinically validated marker of clear-cell renal cell carcinoma (ccRCC) and hypoxic tumors. OncoCAIX is a new ligand for CAIX.

This is a Phase I, multicenter study in patients with suspected ccRCC to evaluate the safety, dosimetry and biodistribution of 68Ga-OncoCAIX for imaging of ccRCC. In this trial, 68Ga-OncoCAIX is offered to ccRCC patients who already received standard of care imaging and might therefore complement available modalities.

All patients will undergo PET/CT imaging with [68Ga]Ga-OncoCAIX. The principal objective of the study is to evaluate safety and dosimetry of a single administration of [68Ga]Ga-OncoCAIX. In addition, data on the uptake, biodistribution, PK and excretion of [68Ga]Ga-OncoCAIX is collected and technical parameters are evaluated.

Patients are divided into two cohorts:

* Cohort A: 3 female + 3 male patients without visceral or bone metastases, which would interfere with dosimetry evaluation of healthy organs.
* Cohort B: all patients who meet the eligibility criteria (up to 14 patients)

Both cohorts are recruited in parallel, and patients are assigned to the respective cohort based on their disease extent. Whenever possible, patients are enrolled in cohort A, unless they are unsuitable for cohort A, or the required number of patients of a given sex has already been enrolled in cohort A.

All patients will receive a single intravenous bolus administration of [68Ga]Ga-OncoCAIX and biodistribution, PK, and dosimetry of [68Ga]Ga-OncoCAIX will be assessed based on a series of PET/CT scans, blood and urine sampling.

Full dosimetry evaluations will be performed for all patients in cohort A. Additional dosimetry in the other patients may be performed to the extent that it is possible based on their disease burden (i.e., only organs not affected by malignant lesions can be evaluated).

All patients will be assessed for safety. In addition, relative uptake to appropriate reference tissue of [68Ga]Ga-OncoCAIX as well as semiquantitative parameters such as SUVmax/SUVmean/SUVsd, are determined. The correlation of [68Ga]Ga-OncoCAIX uptake with immunopathology staining for CAIX will be evaluated in patients undergoing surgery or tumor biopsy collection. The lesion detection rate will be compared to 18F-FDG-PET/CT in patients who receive this as part of their standard diagnostic workup.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected ccRCC (based on standard diagnostic workup).
2. Requirement for diagnostic imaging or diagnostic imaging recently performed.
3. For female patients: negative serum pregnancy test for women of childbearing potential* (WOCBP). WOCBP must agree to use, from the screening to six months following the study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesterone only or combined hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion or vasectomized partner.
4. For male patients: Subjects able to father children must agree to practice effective contraception for three months starting from the study drug administration.
5. Age ≥ 18
6. ECOG ≤ 1
7. Patient must not have any concomitant infections or active concomitant disease.
8. All acute toxic effects (excluding alopecia and fatigue) of any prior therapy (including surgery, radiation therapy, chemotherapy) must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v. 5.0) Grade ≤ 1.
9. Life expectancy of more than 12 weeks.
10. Ability to undergo imaging study procedures.
11. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
12. Willingness and ability to comply with the scheduled visits, plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Chronically impaired renal function as expressed by creatinine clearance < 60 mL/min or serum creatinine > 1.5 x ULN.
2. Presence of active hepatitis.
3. Presence of significant cardiac disorders (congestive heart failure, NYHA class III-IV, myocardial infarction within one year prior to study entry, uncontrolled hypertension, or arrhythmia).
4. Any concomitant condition which in the opinion of investigators makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol.
5. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 4 weeks of administration of the study drug. Minimally invasive procedures such as biopsies are not considered as exclusion criteria.
6. Serious, non-healing wound, ulcer, or bone fracture.
7. Allergy to study medication or excipients in study medication.
8. Any anti-cancer therapy (e.g. cytotoxic chemotherapy, immunotherapy, radiation, surgery, etc.) within 3 weeks before [68Ga]Ga-OncoCAIX-PET/CT scan.
9. Subject has received, or is scheduled to receive, another investigational medicinal product (IMP) from one month before [68Ga]Ga-OncoCAIX injection to end of study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Cohort A: Dosimetry - Effective dose equivalent (mSv) | Assessed on day 1
  Whole-body effective dose (mSv) following administration of a single dose of [68Ga]Ga-OncoCAIX.
Cohort A: Dosimetry - Effective dose absorbed doses (mGy) | Assessed on day 1
  Absorbed doses (mGy) of normal organs following administration of a single dose of [68Ga]Ga-OncoCAIX.
All patients: Safety (AEs and SAEs) | Throughout the study, until a maximum of 7 days after the administration of the study drug.
  Safety of administration of [68Ga]Ga-OncoCAIX, according to Common Terminology Criteria for Adverse Events (CTCAE v.5.0).

SECONDARY OUTCOMES:
Biodistribution profile: SUVmax | Assessed on day 1
  Uptake of [ 68Ga]Ga-OncoCAIX in tumor lesions and healthy organs in terms of SUVmax
Biodistribution profile: SUVmean | Assessed on day 1
  Uptake of [68Ga]Ga-OncoCAIX in tumor lesions and healthy organs in terms of SUVmean
Biodistribution profile: SUVsd | Assessed on day 1
  Uptake of [68Ga]Ga-OncoCAIX in tumor lesions and healthy organs in terms of SUVsd
Pharmacokinetics (PK) - Blood | Assessed on day 1
  Pharmacokinetics (PK) of [68Ga]Ga-OncoCAIX based on measurement on blood of residual radioactivity over time [kBq/mL].
Excretion - Urine | Assessed on day 1
  Excretion of [68Ga]Ga-OncoCAIX based on measurement of residual radioactivity in the urine over time [kBq]

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - ASST Papa Giovanni XXIII, Bergamo, BG
  - IRCCS Ospedale San Raffaele, Milan, Milano
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Milano

IPD SHARING:
Plan to Share IPD: No